CLINICAL TRIAL: NCT06625489
Title: A Phase 1, Randomized, Placebo-Controlled, Double-Blind, Parallel Group Study to Evaluate the Safety, Tolerability and Pharmacokinetics of GSK3915393 Administered as a Single Dose to Healthy Participants of Chinese, Japanese and European Ancestry, and to Assess the Effects of GSK3915393, on the Pharmacokinetics of Nintedanib
Brief Title: A Study to Evaluate the Safety, Tolerability and Blood Levels of GSK3915393 Administered to Healthy Participants of Chinese, Japanese and European Ancestry and to Assess Effects of GSK3915393 on Nintedanib
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 222308
Record Dates: First submitted 2024-10-01; First posted 2024-10-03 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: GSK3915393; Nintedanib; Drug-drug interaction; P-gp inhibitor; Idiopathic pulmonary fibrosis; Interstitial lung disease; Japanese; Chinese; European
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Lung Diseases, Interstitial | interventions — nintedanib

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Part A is a double-blind study and Part B is an open-label study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part A: GSK3915393 (Experimental): Participants from Chinese, Japanese, and European ancestries will be randomized to receive GSK3915393 under fasting condition.
  Interventions: Drug: GSK3915393
- Part A: Placebo (Placebo Comparator): Participants from Chinese, Japanese, and European ancestries will be randomized to receive placebo under fasting condition.
  Interventions: Drug: Part A: Placebo
- Part B: Nintedanib followed by Nintedanib plus GSK3915393 (Experimental): Male participants will be randomized to receive Nintedanib in Period 1 followed by co-administration of Nintedanib and GSK3915393 in Period 2 under fed conditions. There will be a washout period of minimum 5 days post last dose between Period 1 and Period 2.
  Interventions: Drug: Nintedanib; Drug: GSK3915393
- Part B: Nintedanib plus GSK3915393 followed by Nintedanib (Experimental): Male participants will be randomized to receive co-administration of Nintedanib and GSK3915393 in Period 1 followed by Nintedanib in Period 2 under fed conditions. There will be a washout period of minimum 5 days post last dose between Period 1 and Period 2.
  Interventions: Drug: Nintedanib; Drug: GSK3915393

INTERVENTIONS:
Drug: Part A: Placebo — Placebo will be administered.
  Arms: Part A: Placebo
Drug: Nintedanib — Nintedanib will be administered.
  Arms: Part B: Nintedanib followed by Nintedanib plus GSK3915393; Part B: Nintedanib plus GSK3915393 followed by Nintedanib
Drug: GSK3915393 — GSK3915393 will be administered.
  Arms: Part A: GSK3915393; Part B: Nintedanib followed by Nintedanib plus GSK3915393; Part B: Nintedanib plus GSK3915393 followed by Nintedanib

SUMMARY:
GSK3915393 is a new medicine which is being developed for a chronic lung disease called Idiopathic Pulmonary Fibrosis (IPF). This is a healthy participant study which has two parts. Part A will assess the safety, tolerability, and blood levels of GSK3915393 given as a single dose to healthy participants of Chinese, Japanese, and European ancestries. Part B is a drug-drug interaction (DDI) study that examines the effect of a single dose of GSK3915393 on the blood levels of a single dose of nintedanib, which is an approved drug for IPF.

ELIGIBILITY:
Inclusion Criteria:

For Part A and Part B:

Participants who are generally healthy as determined by medical evaluation based on screening medical history, physical examination, vital signs, electrocardiogram (ECG) assessments, and laboratory tests Body weight at least 50.0 kilograms (kg) (110 pounds [lbs]) for male participants (Part A and Part B) or at least 45.0 kg (99 lbs) for female participants (Part A only) Body mass index (BMI) within the range of 18.0 to 28.0 kilogram per square meter (kg/m^2) (inclusive) Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF)

For Part A:

Female Participants: A female participant is eligible to participate if she is not pregnant or breastfeeding, and at least one of the following conditions applies:

Is a woman of non-childbearing potential (WONCBP) Is a woman of childbearing potential (WOCBP) and using an acceptable contraceptive method prior to and during the study intervention period (at a minimum until after the last dose of study intervention). The investigator should evaluate the potential for contraceptive method failure (for example, noncompliance, recently initiated in relationship to the first dose of study intervention) A WOCBP must have a negative highly sensitive pregnancy test within 30 days before the first dose of study intervention Participants of Chinese ancestry are eligible if born in mainland China, Hong Kong or Taiwan; descendant of four ethnic Chinese grandparents and two ethnic Chinese parents; and have lived outside China, Hong Kong or Taiwan for less than 10 years at the time of screening Participants of Japanese ancestry are eligible if born in Japan; Descendant of four ethnic Japanese grandparents and two ethnic Japanese parents; and have lived outside Japan for less than 10 years at the time of screening Participants of European ancestry are eligible if Self-identified as being of European ancestry (i.e. from the original peoples of Europe) irrespective of current place of residence; and descendant of four grandparents and two parents of European ancestry

Exclusion Criteria:

History or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study intervention or interfering with the interpretation of data Participants with systolic blood pressure (BP) greater than (>) 140 millimeter of mercury (mmHg) or diastolic BP > 90 mmHg at screening or pulse rate outside the range of 40 to 100 beats per minute (bpm) will be excluded from the study Alanine transaminase (ALT) or aspartate aminotransferase (AST) >1× upper limit of normal (ULN) Total bilirubin >1.5×ULN; Participants with Gilbert's syndrome can be included with total bilirubin >1.5×ULN as long as direct bilirubin is less than or equal to (≤) 1.5×ULN Current or chronic history of liver disease or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones) QT interval corrected (QTc) >450 milliseconds (msec) at Screening visit based on the average of triplicate ECGs Unable to refrain from the use of prescription or non-prescription drugs, including vitamins, probiotics, antacids, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study intervention, unless in the opinion of the Investigator and the Medical Monitor, the medication will not interfere with the study procedures or compromise participant safety

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2024-10-07 (Actual); Primary Completion 2024-11-25 (Actual); Study Completion 2024-11-25 (Actual)

PRIMARY OUTCOMES:
Part A: Number of Participants with Adverse Events (AEs) | Up to Day 10
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention.
Part A: Number of Participants with Serious Adverse Events (SAEs) | Up to Day 10
  An SAE is defined as any untoward medical occurrence that, at any dose, meets one or more of the criteria: results in death; is life threatening; requires hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect in the offspring of a study participant; abnormal pregnancy outcome; or is a suspected transmission of any infectious agent via an authorized medicinal product.
Part A: Number of Participants with Clinically Significant Changes in Clinical Laboratory Values | Up to Day 10
  Number of participants with clinically significant changes in clinical laboratory values (hematology, clinical chemistry, and routine urinalysis) will be assessed.
Part A: Number of Participants with Clinically Significant Changes in Vital Signs | Up to Day 10
  Number of participants with clinically significant changes in Vital signs (temperature, systolic and diastolic blood pressure [BP], pulse rate and respiratory rate [RR]) will be assessed.
Part A: Number of Participants with Clinically Significant Changes in 12-Lead Electrocardiogram (ECG) | Up to Day 10
  Number of participants with clinically significant changes in 12-lead ECG will be assessed.
Part A: Area Under the Plasma Concentration Versus Time Curve From Time Zero To t (AUC [0-t]) of GSK3915393 | Up to 36 hours post dose
  Blood sample will be collected to evaluate plasma concentration of GSK3915393.
Part A: Area Under the Plasma Concentration Versus Time Curve From Time Zero To Infinity (AUC [0-inf]) of GSK3915393 | Up to 36 hours post dose
  Blood sample will be collected to evaluate plasma concentration of GSK3915393.
Part A: Maximum Observed Plasma Concentration (Cmax) of GSK3915393 | Up to 36 hours post dose
  Blood sample will be collected to evaluate plasma concentration of GSK3915393.
Part A: Time to Cmax (Tmax) of GSK3915393 | Up to 36 hours post dose
  Blood sample will be collected to evaluate time of maximum plasma concentration of GSK3915393.
Part A: Apparent Terminal Half-life (T1/2) of GSK3915393 | Up to 36 hours post dose
  Blood sample will be collected to evaluate plasma concentration of GSK3915393.
Part B: AUC (0-t) of Nintedanib | Up to 48 hours post dose
  Blood sample will be collected to evaluate plasma concentration of Nintedanib.
Part B: AUC (0-inf) of Nintedanib | Up to 48 hours post dose
  Blood sample will be collected to evaluate plasma concentration of Nintedanib.
Part B: Cmax of Nintedanib | Up to 48 hours post dose
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention

SECONDARY OUTCOMES:
Part B: Number of Participants with AEs | Up to Day 17
  An SAE is defined as any untoward medical occurrence that, at any dose, meets one or more of the criteria: results in death; is life threatening; requires hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect in the offspring of a study participant; abnormal pregnancy outcome; or is a suspected transmission of any infectious agent via an authorized medicinal product.
Part B: Number of Participants with SAEs | Up to Day 17
  Number of participants with clinically significant changes in clinical laboratory values (hematology, clinical chemistry, and routine urinalysis) will be assessed.
Part B: Number of Participants with Clinically Significant Changes in Clinically Laboratory Values | Up to Day 17
  Number of participants with clinically significant changes in vital signs (temperature, systolic and diastolic BP, pulse rate and RR) will be assessed.
Part B: Number of Participants with Clinically Significant Changes in Vital Signs | Up to Day 17
  Number of participants with clinically significant changes in 12-lead ECG will be assessed.
Part B: Number of Participants with Clinically Significant Changes in 12-Lead ECG | Up to Day 17
  Blood sample will be collected to evaluate the time of maximum plasma concentration of Nintedanib.
Part B: Tmax of Nintedanib | Up to 48 hours post dose
  Blood sample will be collected to evaluate plasma concentration of Nintedanib.
Part B: T1/2 of Nintedanib | Up to 48 hours post dose

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - GSK Investigational Site, Cypress, California
  - GSK Investigational Site, Las Vegas, Nevada

IPD SHARING:
Plan to Share IPD: Yes
GSK will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or asset(s) with development terminated across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months, but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/